CLINICAL TRIAL: NCT02196961
Title: Prospective Randomized Trial of an Adjuvant Therapy of Completely Resected Merkel Cell Carcinoma (MCC) With Immune Checkpoint Blocking Antibodies (Nivolumab, Opdivo®; Ipilimumab (Yervoy®) Every 3 Weeks for 12 Weeks Versus Observation
Brief Title: Adjuvant Therapy of Completely Resected Merkel Cell Carcinoma With Immune Checkpoint Blocking Antibodies vs Observation
Acronym: ADMEC-O
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. med. Dirk Schadendorf (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dirk Schadendorf, Prof. Dr. med. Dirk Schadendorf, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-205
Record Dates: First submitted 2014-06-20; First posted 2014-07-22 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Merkel Cell Carcinoma
Keywords: Merkel cell carcinoma; Adjuvant; Nivolumab
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): After complete resection of Merkel cell carcinoma, patients randomized to the observational arm will be observed only
- Nivolumab (Experimental): After complete resection of Merkel cell carcinoma, patients randomized to the treatment arm will receive nivolumab at a fixed dose of 480 mg by IV infusion every 4 weeks for up to one year (i.e.13 doses).
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — adjuvant treatment of completely resected Merkel cell carcinoma
  Other Names: Opdivo
  Arms: Nivolumab

SUMMARY:
Primary objective: To estimate the efficacy of adjuvant nivolumab monotherapy in completely resected MCC patients

Primary endpoint: Disease-free survival (DFS) rate evaluated at 12, 24 and 48 months after date of randomization

Secondary Objectives: To describe the safety profile and additional efficacy parameters of the nivolumab treatment in MCC

Secondary endpoints:

* Adverse events according to CTCAE, Version 4.0 criteria, that are related to the administration of nivolumab
* Disease-free survival (DFS)
* Overall survival (OS) and OS rates at 12, 24 and 48 months after randomization

Explorative Endpoints:

* Distant-metastases-free survival (DMFS) and DMFS rate at 12, 24 and 48 months after randomization
* Identification and validation of prognostic/predictive biomarkers
* Quality of life (EORTC QLQ-C30) until 24 months after randomization

DETAILED DESCRIPTION:
This is an international, open-label, randomized, multicenter phase II study to assess the efficacy of adjuvant nivolumab therapy in completely resected MCC patients. In the initial trial design, the immune modulating treatment was based on CTLA-4 blockade by ipilimumab; however, the advent of PD-1/PD-L1 blockade in the palliative treatment of MCC (presented at AACR, ASCO and ESMO) dramatically changed the treatment environment to an extent that applying treatments other than by PD-1/PD-L1 blockade had become very difficult. Moreover, the side effects of PD-1/PD-L1 blocking are far less frequent than side effects of ipilimumab. Consequently, randomization into the previous Ipilimumab treatment arm A was stopped. New patients will be randomized to nivolumab treatment instead. Patients randomized already into the Ipilimumab-arm will be evaluated descriptively for efficacy and safety. Patients already randomized into the observation arm (arm B) will be evaluated together with the newly randomized arm B-patients. A total of 177 patients with completely resected MCC will be enrolled over a recruitment period of 36 months into this trial, and randomized 2:1 as mentioned above. Patients will be stratified by sex, age, and stage of disease.

Examinations and Follow-up Phase:

The disease will be assessed at baseline, and thereafter every 12 weeks according to the current German guidelines for the management of MCC patients for 24 months after randomization, or until withdrawal of informed consent, lost to follow-up, or death, whichever occurs first. In addition, the patient's quality of life will be evaluated at baseline (pretreatment visit) and every 3 months until 24 months after randomization using a standard questionnaire (EORTC QLQC30).

After 24 months, additional FU visits (or phone calls) will be conducted 6-monthly recording survival and tumor status including subsequent therapies until withdrawal of informed consent, lost to follow-up, death or end of study, whichever occurs first.

End of study is defined as 48 months post LPFV (last patient first visit = date of randomization).

Same methods of assessment (e.g. ultrasonography, CT or MRI scans) used at baseline will be used during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing and able to give written informed consent.
2. Central histological confirmation of diagnosis of Merkel cell carcinoma (MCC).
3. All MCC manifestations have been completely resected by surgery within 12 weeks before enrolment.
4. No currently present metastases (as confirmed by standard imaging studies (e.g. suggested by S2k guidelines)).
5. No previous systemic therapy for MCC.
6. Required values for initial laboratory tests:

   * WBC ≥ 2000/uL
   * ANC ≥ 1000/uL
   * Platelets ≥ 75 x 103/uL
   * Hemoglobin ≥ 8 g/dL (≥ 80 g/L)
   * Creatinine ≤ 2.0 x ULN
   * AST/ALT ≤ 2.5 x ULN
   * Total Bilirubin ≤ 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
7. ECOG performance status 0 or 1.
8. No active or chronic infection with HIV, Hepatitis B (HBV) or C (HCV).
9. Men and women, ≥ 18 years of age.
10. Women of childbearing potential (WOCBP) must be using an adequate method of contraception (Pearl-Index < 1) to avoid pregnancy during treatment phase and for additional 5 months after the last dose of nivolumab, in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of nivolumab.
11. Men of fathering potential must be using an adequate method of contraception to avoid conception and for 7 months after the last dose of nivolumab in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

1. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease requiring systemic steroids (e.g., rheumatoid arthritis, systemic progressive sclerosis, systemic lupus erythematosus, autoimmune vasculitis); autoimmune motor neuropathy.
2. Other serious illnesses, e.g., serious infections requiring i.v. antibiotics.
3. The patient is known to be positive for Human Immunodeficiency Virus (HIV) or other chronic infections (HBV, HCV) or has another confirmed or suspected immunosuppressive or immune deficient condition.
4. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of nivolumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea.
5. Any non-oncology vaccine therapy for up to 1 month before or after any dose of nivolumab.
6. A history of prior or current treatment with a T cell potentiating agent (e.g. IL-2, interferon, anti-CTLA-4, anti-CD137, anti-PD1, anti-PD-L1, or anti-OX40 antibody).
7. Chronic use of immunosuppressive agents or systemic corticosteroids.
8. Women of childbearing potential (WOCBP), defined above in Section 5.1, who:

   * are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for additional 5 months after the last dose of investigational product
   * have a positive pregnancy test at baseline
   * are pregnant or breastfeeding.
9. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
10. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.
11. Men of reproductive potential unwilling to use an adequate method to avoid pregnancy for additional 7 months after the last dose of investigational product.
12. Use of any investigational or non-registered product (drug or vaccine) other than the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) rate at 12 months | 1 years post last patient first treatment/randomization
  The number of patients alive and free of disease at 12 months after randomization in arm A compared to DFS in arm B.
Disease-free survival (DFS) rate at 24 months | 2 years post last patient first treatment/randomization
  The number of patients alive and free of disease at 24 months after randomization
Disease-free survival (DFS) rate at 48 months | 4 years post last patient first treatment/randomization
  The number of patients alive and free of disease at 48 months after randomization

SECONDARY OUTCOMES:
Number of adverse events | 1, 2 and 4 years post last patient first treatment/randomization
  Adverse events according to CTCAE, Version 4.0 criteria, that are related to the administration of Ipilimumab
Overall survival rate at 12 months | 1 year post last patient first treatment/randomization
  Overall survival rate at 12 months, defined as the number of patients alive at 12 months after randomization divided by the total number of patients randomized.
Overall survival rate at 24 months | 2 years post last patient first treatment/randomization
  Overall survival rate at 24 months, defined as the number of patients alive at 24 months after randomization divided by the total number of patients randomized.
Overall survival rate at 48 months | 4 years post last patient first treatment/randomization
  Overall survival rate at 48 months, defined as the number of patients alive at 48 months after randomization divided by the total number of patients randomized.
Disease-free survival (DFS) | 1, 2 and 4 years post last patient first treatment/randomization
  Time from randomization to recurrence of tumor
Overall survival (OS) | 1, 2 and 4 years post last patient first treatment/randomization
  Time from randomization to death of patient

OTHER OUTCOMES:
Distant-metastases-free survival (DMFS) at 12 months after randomization | 1 year post last patient first treatment/randomization
  Number of patients free of distant metastases at 12 months after randomization
Distant-metastases-free survival (DMFS) at 24 months after randomization | 2 years post last patient first treatment/randomization
  Number of patients free of distant metastases at 24 months after randomization
Distant-metastases-free survival (DMFS) at 48 months after randomization | 4 years post last patient first treatment/randomization
  Number of patients free of distant metastases at 48 months after randomization
Identification of prognostic/predictive biomarkers | 2 and 4 years post last patient first treatment/randomization
  Identify and validate prognostic/predictive biomarkers such as immune status, kinetics of the absolute lymphocyte count (ALC), or tumor microenvironment characteristics
Quality of life (EORTC QLQ-C30) until 24 months after randomization | 2 years post last patient first treatment/randomization
  The patient's quality of life will be evaluated at baseline (pretreatment visit) and every 3 months until 24 months after randomization using a standard questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (20):
- Germany (19):
  - University Hospital Essen, Dermatology, Essen, North Rhine-Westphalia
  - Charité Universitätsmedizin Berlin, Berlin
  - Elbeklinikum Buxtehude, Buxtehude
  - University Hospital Dresden, Dermatology, Dresden
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - SRH Wald-Klinikum Gera, Gera
  - Hannover Medical School, Hanover
  - National Centre for Tumour Diseases (NCT), Heidelberg
  - University Hospital Schleswig-Holstein, Kiel, Kiel
  - Universitätsklinikum Leipzig Klinik u. Poliklinik f. Dermatologie, Venerologie u. Allergologie, Leipzig
  - Universitätsklinikum Mainz Hautklinik und Poliklinik, Mainz
  - Universitätsklinikum Mannheim Klinik f. Dermatologie, Venerologie u. Allergologie, Mannheim
  - University Hospital München (LMU), Munich
  - Universitätsklinikum Münster Zentrale Studienkoordination für innovative Dermatologie (ZID), Münster
  - Specialist clinic in Hornheide, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - University Hospital Tübingen, Tübingen
  - Universitätsklinikum Würzburg Klinik u. Poliklinik f. Dermatologie, Venerologie u. Allergologie, Würzburg
- The Netherlands Cancer Institute / Antoni van Leeuwenhoek Hospital (NKI/AVL), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becker JC, Ugurel S, Leiter U, Meier F, Gutzmer R, Haferkamp S, Zimmer L, Livingstone E, Eigentler TK, Hauschild A, Kiecker F, Hassel JC, Mohr P, Fluck M, Thomas I, Garzarolli M, Grimmelmann I, Drexler K, Spillner AN, Eckhardt S, Schadendorf D; DeCOG. Adjuvant immunotherapy with nivolumab versus observation in completely resected Merkel cell carcinoma (ADMEC-O): disease-free survival results from a randomised, open-label, phase 2 trial. Lancet. 2023 Sep 2;402(10404):798-808. doi: 10.1016/S0140-6736(23)00769-9. Epub 2023 Jul 11. PMID 37451295